CLINICAL TRIAL: NCT07042737
Title: The Effect of Education Provided to Women in Menopause Through Animation on Breast Cancer Attitudes, Behaviors, and Screening Test Participation
Brief Title: The Effect of Animation-Based Education on Menopausal Women's Attitudes, Behaviors, and Screening Test Participation Regarding Breast Cancer
Acronym: Menopause
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Simge Ozturk, principal ınvestigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Inonu7
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Menopausal Women; Education Nursing; Breast Cancer Females; Motivation; Screening Strategy
Keywords: education through animation; menopause; breast cancer; screening test; motivation
MeSH Terms: conditions — Breast Neoplasms | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Participants identified by researchers prior to the start of the study were divided into experimental and control groups using a randomization method. Women in the experimental group will receive 40-45 minute training sessions once a week for one week on specified days and times. The training sessions will be conducted in groups of 8-12 people. The content of the training sessions will include information about the purpose, duration, and rules of the training. After the information is provided, a pre-test will be administered. Using the face-to-face interview method, researchers involved in the study will show animated videos enriched with sound and images through an online program they have prepared, lasting 10-12 minutes. A mid-test will be conducted 14 days after the pre-test. Three months after the pre-test, the women participating in the study will be contacted, and a final test will be administered in their own homes.
Who Masked: Investigator, Outcomes Assessor
Masking Description: After randomization was performed by an independent researcher, the experimental group and control group were determined by lottery. In addition, the data will be analyzed by S.Ö., a researcher who did not collect the data, using masked data. The experimental and control groups will be assigned as A and B in the analysis program in such a way that S.Ö. will not know which group is which.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group: Breast cancer education group through animation (Experimental): The experimental group, determined by random selection, will include 68 women in menopause. These women will be asked to give their consent to participate in the study. After consent is obtained, a preliminary test will be conducted. Then, women in menopause will be educated on the symptoms and signs of breast cancer based on animation, self-breast examination, clinical breast examination, and mammography. The application will be conducted once a week. An interim test was conducted 14 days after the application, and a final test was conducted three months later.
  Interventions: Behavioral: animation-based breast cancer education
- control group (Sham Comparator): No intervention was applied to the control group.
  Interventions: Other: Control group (placebo)

INTERVENTIONS:
Behavioral: animation-based breast cancer education — The animation-based humorous application consists of four videos, each lasting 40-45 minutes, which separately explain the signs and symptoms of breast cancer, self-breast examination, clinical breast examination, and mammography through animation.
  Arms: experimental group: Breast cancer education group through animation
Other: Control group (placebo) — No intervention will be applied to the control group.
  Arms: control group

SUMMARY:
The aim of this study was to determine the effect of education provided to women in menopause through animation on their attitudes toward breast cancer, behaviors, and screening test participation. The study will include a total of 136 women in the menopausal period, comprising 68 experimental group participants and 68 control group participants who have applied to the Orduyeri and Kırtepe Family Health Centers affiliated with the Bartın Public Health Institution. Women who agree to participate in the project, which will run from January to August 2025, will receive 40-45 minute training sessions in a suitable room at the ASM. The training sessions will be conducted in groups of 8-12 people. The training content will include information about the purpose, duration, and rules of the training. After providing information about the project, a pre-test will be administered. Through face-to-face interviews, researchers assigned to the project will show animated videos enriched with sound and images via an online program they have prepared. These videos will be 10-12 minutes long, and an interim test will be conducted. Three months after the pre-test, the women participating in the study will be contacted, and a final test will be administered in their own homes. Project data will be collected using the Personal Information Form, Champion Health Belief Scale, and Breast Cancer Awareness Scale. Descriptive statistics, independent sample t-tests, chi-square tests, and repeated measures analysis of variance (ANOVA) tests will be used in the statistical analysis of the project.

DETAILED DESCRIPTION:
Menopause is a stage of life in which women's reproductive functions cease due to a decline in ovarian activity and a corresponding decrease in the hormones produced by the ovaries. Seventy percent of women in menopause experience at least one symptom related to menopause. These symptoms can negatively affect women's daily lives, quality of life, interpersonal relationships, and sexual lives. Additionally, it increases women's risk of health issues such as breast cancer, cardiovascular disease, and obesity. Women's perceptions, attitudes, and behaviors toward menopause determine the methods they use to cope with these symptoms and health issues. Women spend one-third of their lives in menopause and use methods such as lifestyle changes, reflexology, massage, acupressure, and listening to music to cope with menopause symptoms and issues. Animation-based education is extremely important in terms of improving the quality of education and ensuring women's self-confidence and focus. There are studies in the literature that examine the effect of educational programs on breast cancer attitudes, behaviors, and screening test status in order to cope with menopausal symptoms and breast cancer. However, no studies have been found that evaluate educational applications delivered through animation, which is thought to increase the effectiveness of education. Based on this, this study was designed to determine the effect of education delivered through animation to women in menopause on breast cancer attitudes, behaviors, and screening test participation. The study will include a total of 136 women in the menopausal period, comprising 68 experimental group participants and 68 control group participants who have applied to the Orduyeri and Kırtepe Family Health Centers affiliated with the Bartın Public Health Institution. Women who agree to participate in the project, which will run from January to August 2025, will receive 40-45 minute training sessions in a suitable room at the ASM. The training sessions will be conducted in groups of 8-12 people. The training content will include information about the purpose, duration, and rules of the training. After providing information about the project, a pre-test will be administered. Through face-to-face interviews, researchers assigned to the project will show animated videos enriched with sound and images via an online program they have prepared. These videos will be 10-12 minutes long, and an interim test will be conducted. Three months after the pre-test, the women participating in the study will be contacted, and a final test will be administered in their own homes. Project data will be collected using the Personal Information Form, Champion Health Belief Scale, and Breast Cancer Awareness Scale. Descriptive statistics, independent sample t-tests, chi-square tests, and repeated measures analysis of variance (ANOVA) tests will be used in the statistical analysis of the project.

ELIGIBILITY:
Inclusion Criteria:

* Not having been diagnosed with breast cancer,
* not performing regular self-examinations (those who performed self-examinations at least once a month were excluded),
* not having had a mammogram (those who had a mammogram within the first six months after training were excluded),
* not having undergone a clinical breast examination (those who underwent a clinical breast examination within the first 6 months after the training were excluded),
* not breastfeeding or being pregnant, being literate, owning a smartphone,
* having internet access,
* not having uterine abnormalities,
* having ovaries,
* not having used sex hormones.

Exclusion Criteria:

* never experiencing menopausal symptoms,
* undergoing surgical menopause,
* currently or previously using hormonal therapy,
* having a psychiatric disorder,
* having menstruated in the past year,
* incomplete forms,
* not fully participating in video-based education programs.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — women going through menopause
Enrollment: 136 (Estimated)
Dates: Start 2025-06-20 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-10-20 (Estimated)

PRIMARY OUTCOMES:
menopause symptom scale | 3 month
  The scale consists of a total of 11 items and 3 subscales. These 3 subscales are called the "Somatic Complaints subscale," "Psychological Complaints subscale," and "Urogenital Complaints subscale." The scale is a 5-point Likert scale. The score obtained from the scale ranges from 0 to 44 points. An increase in the total score obtained from the scale indicates an increase in the severity of menopausal complaints experienced.

SECONDARY OUTCOMES:
Champion Health Belief Model Scale | 3 month
  The scale has eight subscales and consists of 58 items. These are: importance/seriousness, sensitivity, health motivation, benefits and barriers to self-breast examination, self-efficacy, and benefits and barriers to mammography. Scale items are scored on a scale of 1 to 5. The lowest score for all dimensions of the scale is the sum of the lowest scores of the subgroup, and the highest score is the sum of the highest scores of the subgroup. It has been noted that as the score obtained from the scale increases, the subdimensions also increase.
Breast Cancer Awareness Scale | 3 month
  The scale consists of a total of 13 items, including symptoms (11 items), breast examination frequency (1 item), and age of breast cancer (1 item), to determine the breast cancer awareness scale. There is no cut-off point for the scale. When 5 symptoms are reported, 1 point is awarded; when a woman aged 70 is indicated, 1 point is awarded; and when a monthly breast examination is reported, 1 point is awarded. Incorrect answers receive 0 points. Scoring ranges from 0 to 3. It has been determined that as the score from the scale increases, breast cancer awareness also increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu University, Bartın, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No